CLINICAL TRIAL: NCT04651816
Title: Penn State Health (PSH) Diabetes Prevention Program (DPP) Pilot
Brief Title: Diabetes Prevention Program Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Dennis P. Scanlon, Distinguished Professor of Health Policy and Administration, Director of the Center for Health Care and Policy Research, Penn State University
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 00010222
Record Dates: First submitted 2020-11-24; First posted 2020-12-03 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-09

CONDITIONS: Pre-diabetes
MeSH Terms: conditions — Glucose Intolerance

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not know what intervention group they will be assigned to (motivational messaging, incentives or control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control PSH DPP only (Active Comparator): This group will be enrolled the PSH DPP program. There will be two cohorts for this arm.
  Interventions: Behavioral: DPP Program
- Treatment 1 Financial Incentives A (Experimental): This group will receive gift cards as financial incentive to participate in the PSH DPP program. There will be two cohorts for this arm.
  Interventions: Behavioral: Financial Incentives; Behavioral: DPP Program
- Treatment 2 Financial Incentives B (Experimental): This group will receive gift cards as financial incentive to participate in the PSH DPP program. There will be two cohorts for this arm.
  Interventions: Behavioral: Financial Incentives; Behavioral: DPP Program
- Treatment 3 Motivational Text Messaging (Experimental): This group will receive text messages with motivational messages while participating in the PSH DPP program. There will be two cohorts for this arm.
  Interventions: Behavioral: Motivational Message; Behavioral: DPP Program

INTERVENTIONS:
Behavioral: Financial Incentives — Participants will be entered into a lottery to receive a gift card for class attendance.
  Arms: Treatment 1 Financial Incentives A; Treatment 2 Financial Incentives B
Behavioral: Motivational Message — Participants will be sent motivational messages through out their participation in the PSH DPP program.
  Arms: Treatment 3 Motivational Text Messaging
Behavioral: DPP Program — All Participants will be enrolled in the DPP program.

SUMMARY:
This initiative, which is a partnership between State College area Penn State Health ambulatory care clinics located off campus in the State College area, has two primary goals: 1) improve the health and quality of life of Penn State Health patients with pre-diabetes and 2) decrease associated health care costs due to type 2 diabetes and its complications. The results from the study may serve as a model for additional chronic disease prevention programs to implement in additional Penn State Health clinics in the future.

DETAILED DESCRIPTION:
Through this initiative, providers in Penn State Health ambulatory health care clinics (PSH clinics) will identify pre-diabetic patients to take part in a Diabetes Prevention Program (DPP), modeled after the Centers for Disease Control's (CDC) program.

The DPP is a CDC-recognized lifestyle change program developed specifically to prevent type 2 diabetes. It is designed for people who have prediabetes or are at risk for type 2 diabetes, but who do not already have diabetes. We will be using the DPP distance learning program which allows online delivery of classes. A trained lifestyle coach leads the program to help subjects change certain aspects of their lifestyle, like eating healthier, reducing stress, and getting more physically activity. The program also includes group support. The DPP is a year-long program focused on long-term changes and lasting results. Key components of the program include a CDC-approved curriculum with lessons, handouts, and other resources; a lifestyle coach, specifically trained to lead the program; and a support group of people with similar goals and challenges.

To that end, this study has multiple arms that will test whether participation in the PSH DPP - and exposure to motivational messages that encourage physical activity or participation in lotteries, an increasingly common strategy for behavioral motivation, - significantly improves program retention and health-related outcomes, compared to those who only participate in the PSH DPP.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years old and under age 65 AND
2. Body Mass Index ≥25 kg/m2 (≥23 kg/m2 if Asian) AND
3. Not be pregnant at time of enrollment AND
4. Have no previous diagnosis of type 1 or type 2 diabetes AND
5. Have a blood test result in the prediabetes range within the past year, meeting one of these specifications:

   1. Hemoglobin A1c: 5.7-6.4%, OR
   2. Fasting plasma glucose : 100-125 mg/dL, OR
   3. Two-hour plasma glucose (after a 75-gm glucose load): 140-199 mg/dL, OR
   4. Have a previous clinical diagnosis of gestational diabetes mellitus (GDM), AND
6. Not in hypertensive crisis with systolic over 180 and/or diastolic over 120
7. Be an established patient at a Penn State Health clinic in State College, PA (i.e. have at least one visit in past 18 months) AND
8. Fluent in English AND
9. Own and carry an iPhone (running iOS version 10 or higher) or Android (running operating system 7 or higher) smartphone during waking hours
10. Internet access
11. Tablet or desktop/laptop computer with webcam for classes
12. Active email address

Exclusion Criteria:

1. Under 18 years old and over age 65
2. Body Mass Index <25 kg/m2 (<23 kg/m2 if Asian)
3. Pregnant at the time of enrollment
4. Previous diagnosis of type 1 or type 2 diabetes
5. Have a blood test result within the past year meeting one of these specifications:

   1. Hemoglobin A1c: not in range of 5.7-6.4%
   2. Fasting plasma glucose: not in range of 100-125 mg/dL
   3. Two-hour plasma glucose (after a 75-gm glucose load): not in range of 140-199 mg/dL
   4. No previous clinical diagnosis of gestational diabetes
6. Active hypertensive crisis with systolic over 180 and/or diastolic over 120 (patients in this category would be referred to primary care provider for immediate visit)
7. Not be an established patient at a Penn State Health clinic in State College, PA (i.e. have not had at least one visit in the past 18 months)
8. Not fluent in English
9. Not own and carry an iPhone (running iOS version 10 or higher) or Android (running operating system 7 or higher) smartphone during waking hours.
10. Decisional impairment
11. Prisoner status
12. Actively taking any of the following drug classes: Biguanides, Sulfonylureas (SU), Thiazolidendiones (TZD), Meglitinides, Alpha-glucosidase inhibitors, Dipetidyl Peptidase-IV (DPP4) inhibitors, Insulin , Sodiumglucose transporter 2 (SGLT2) inhibitors, glucagon-like peptide-1 (GLP-1) .
13. Anyone who does not have internet access
14. Anyone who does not have tablet or desktop/laptop computer with webcam
15. Anyone who does not have an active email address

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-08-08 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Weight Loss | 12 months
  Patients will be monitored through out the study for healthy weight loss.
Subject Retention | 12 months
  Participants will be tracked for retention throughout the study.

SECONDARY OUTCOMES:
Blood Pressure | 12 months
  Participant blood pressure will be monitored through out the study for change.
A1c | 12 months
  Participant A1c will be monitored through out the study for change.
Total Cholesterol | 12 months
  Participant total cholesterol will be monitored through out the study for change.
Pregnancy Status | 12 months
  Participant pregnancy status will be reported throughout the study if status changes from baseline.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | 12 months
  Participants will complete the KOOS survey as part of this study.
Quality of Life (SF-36) | 12 months
  Participants will complete the SF-36 as part of this study.
Opinions about PSH DPP program | 12 months
  Participants will provide feedback and opinions about the PSH DPP program via survey at the conclusion of the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Health Medical Group -- Park Avenue, State College, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Do to be determined.